CLINICAL TRIAL: NCT05372315
Title: A Randomized, Controlled Study to Evaluate the Safety and Effectiveness of Treatment With an Intracanalicular Dexamethasone (0.4mg) Ophthalmic Insert in the Operating Room Following Cataract Surgery/Intraocular Lens Implant (IOL).
Brief Title: Efficacy of Dextenza Insert in Upper vs Lower Punctum Following Cataract Surgery With PCIOL.
Acronym: DEXTENZA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Iworks Laser and Vision Center (Other)
Collaborators: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Patrick Spencer, Principal Investigator, Iworks Laser and Vision Center
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SPENCER-2022-401
Record Dates: First submitted 2022-05-06; First posted 2022-05-12 (Actual); Results first posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-07

CONDITIONS: Cataract
Keywords: PCIOL; CCI CE
MeSH Terms: conditions — Cataract | interventions — Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: Each subject's participation is expected to last for approximately 1 month and will be required to complete six scheduled visits over the course of the study period: Baseline (Screening Visit), Operative Visit/Insertion Day (Day 0), Day 1, Day 8, Day 14 and Day 30.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lower Punctum Insertion (Group 1) (Other): DEXTENZA (dexamethasone ophthalmic insert, 0.4mg) for intracanalicular use
  Group 1 (up to 40 eyes) will receive the insert in the lower punctum on the day of surgery in the OR.
  Interventions: Drug: Dextenza 0.4Mg Ophthalmic Insert
- Upper Punctum Insertion (Group 2) (Other): DEXTENZA (dexamethasone ophthalmic insert, 0.4mg) for intracanalicular use
  Group 2 (up to 40 eyes) will receive the insert in the upper punctum on the of surgery in the OR.
  Interventions: Drug: Dextenza 0.4Mg Ophthalmic Insert

INTERVENTIONS:
Drug: Dextenza 0.4Mg Ophthalmic Insert — (dexamethasone ophthalmic insert)-for the treatment of ocular inflammation and pain following following ophthalmic surgery.

SUMMARY:
To assess the safety and effectiveness of treatment with an intracanalicular dexamethasone (0.4mg) insert in the operating room following cataract surgery/intraocular lens implant (IOL) with or without iStent/Hydrus/Goniotomy when placed in the lower punctum compared to the upper punctum.

DETAILED DESCRIPTION:
This is a randomized, controlled study to evaluate the safety and effectiveness of treatment with an intracanalicular dexamethasone (0.4mg) insert in the operating room following cataract surgery/intraocular lens implant (IOL) with or without iStent/Hydrus/Goniotomy when placed in the lower punctum compared to the upper punctum.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for study participation if they:

1. Are planning to undergo non-complicated CCI CE/PCIOL in one or both eyes with or without iStent/Hydrus/Goniotomy.
2. Are willing and able to comply with clinic visits and study related procedures.
3. Are willing and able to sign the informed consent form.
4. Not pregnant.

Exclusion Criteria:

Subjects are not eligible for study participation if they:

1. Are currently being treated with corticosteroid implant (i.e. Ozurdex).
2. Have a history of herpes simplex virus keratitis or present active bacterial, viral, or fungal keratitis in either eye.
3. Have a history of complete punctal occlusion in one or both punctum.
4. Currently use topical ophthalmic steroid medications.
5. Are unwilling or unable to comply with the study protocol.
6. Are determined by the Investigator to not be included for reasons not already specified (e.g., systemic, behavioral, or other ocular disease/abnormality) or if the health of the subject or the validity of the study outcomes may be compromised by the subject's enrollment.
7. Have active infectious systemic disease.
8. Have active infectious ocular or extraocular disease.
9. Have unobstructed nasolacrimal duct in the study eye(s) (dacrocystitis).
10. Have known hypersensitivity to dexamethasone or are a known steroid responder.
11. Have a history of ocular inflammation or macular edema.
12. Are currently being treated with immunomodulating agents in the study eye(s).
13. Are currently being treated with immunosuppressants an/or oral steroids.
14. Are Pregnant or breast-feeding or wish to become pregnant during the length of study participation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick L Spencer, DO, Principal Investigator — Iworks Laser & Vision Center
Locations (1):
- Iworks Laser & Vision Center, Dayton, Ohio, United States

REFERENCES:
- [Background] Greenwood MD, Gorham RA, Boever KR. A Randomized Fellow-Eye Clinical Trial to Evaluate Patient Preference for Dexamethasone Intracanalicular Insert or Topical Prednisolone Acetate for Control of Postoperative Symptoms Following Bilateral Femtosecond Laser in Site Keratomileusis (LASIK). Clin Ophthalmol. 2020 Aug 6;14:2223-2228. doi: 10.2147/OPTH.S265311. eCollection 2020. PMID 32821083

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single medical clinic open enrollment from June-October 2022.
Groups:
- Lower Punctum Insertion (Group 1); Upper Punctum Insertion (Group 2): Participants undergoing cataract surgery with IOL implant with or with out Istent, Hydrus, or Goniotomy who will receive dexamethasone ophthalmic insert 0.4mg).
Period: Overall Study
Arm/Group | Lower Punctum Insertion (Group 1) | Upper Punctum Insertion (Group 2)
Started | 40 | 40
Completed | 39 | 40
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lower Punctum Insertion (Group 1): DEXTENZA (dexamethasone ophthalmic insert, 0.4mg) for intracanalicular use
  Group 1 (up to 40 eyes) will receive the insert in the lower punctum on the day of surgery in the OR.
  Dextenza 0.4Mg Ophthalmic Insert: (dexamethasone ophthalmic insert)-for the treatment of ocular inflammation and pain following following ophthalmic surgery, and ocular itching associated with allergic conjunctivitis.
- Upper Punctum Insertion (Group 2): DEXTENZA (dexamethasone ophthalmic insert, 0.4mg) for intracanalicular use
  Group 2 (up to 40 eyes) will receive the insert in the upper punctum on the of surgery in the OR.
  Dextenza 0.4Mg Ophthalmic Insert: (dexamethasone ophthalmic insert)-for the treatment of ocular inflammation and pain following following ophthalmic surgery, and ocular itching associated with allergic conjunctivitis.
- Total: Total of all reporting groups
Arm/Group | Lower Punctum Insertion (Group 1) | Upper Punctum Insertion (Group 2) | Total
Number analyzed (Participants) | 39 | 40 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] — Age range 18-100 years old.
  years | 68.5 (8.1) | 68.3 (9.1) | 68.4 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 26 | 49
  Male | 16 | 14 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 4 | 6 | 10
  Race: African American | 35 | 34 | 69
Surgical Procedure [Count of Participants; unit: Participants]
  Cataract Surgery Only | 35 | 35 | 70
  Cataract-MIGS | 4 | 5 | 9
Cataract Type [Count of Participants; unit: Participants]
  Nuclear | 27 | 26 | 53
  Cortical | 12 | 14 | 26

OUTCOME MEASURES:

1. Primary Outcome: Participants With Complete Absence of Ocular Pain at Day 8
Description: Participant reported ocular pain on a scale of (0-10) with zero (0) equaling no pain and ten(10) equaling maximal pain on day 8.
Time Frame: at Day 8
Population: Participants with complete absence of ocular pain at day 8
Measure: Count of Participants; unit: Participants
Groups:
- Lower Punctum Insertion (Group 1); Lower Punctum Insertion (Group 2): Dexamethasone ophthalmic insert, 0.4mg intracanalicular insert in the lower punctum on the day of surgery in the OR.
Arm/Group | Lower Punctum Insertion (Group 1) | Lower Punctum Insertion (Group 2)
Number analyzed (Participants) | 39 | 40
Participants
  No Post Op Pain Reported | 39 | 39
  Post Op Pain Reported | 0 | 1

2. Primary Outcome: Participants With Zero Cells on Day 14
Description: Proportion of of participants with complete absence of anterior chamber cell at Day 14 as measured by Summed Ocular Inflammation Score (0-4).
Time Frame: at Day 14
Population: Lower and Upper Punctum Insertion
Measure: Count of Participants; unit: Participants
Groups:
- Upper Punctum Insertion (Group 2): Dexamethasone ophthalmic insert, 0.4mg intracanalicular insert in the lower punctum on the day of surgery in the OR.
Arm/Group | Lower Punctum Insertion (Group 1) | Upper Punctum Insertion (Group 2)
Number analyzed (Participants) | 39 | 40
Participants
  Patients with Zero Cell | 38 | 37
  Patients with Cell | 1 | 3

3. Secondary Outcome: Ease of Insertion
Description: Rated as Easy, Moderate, Difficult
Time Frame: Day 0
Population: Easy, Moderate, Difficult.
Measure: Count of Participants; unit: Participants
Arm/Group | Lower Punctum Insertion (Group 1) | Upper Punctum Insertion (Group 2)
Number analyzed (Participants) | 39 | 40
Participants
  Easy | 36 | 36
  Moderate | 2 | 4
  Difficult | 1 | 0

4. Secondary Outcome: Attempts to Achieve Successful Insertion
Description: Number of attempts to insert the dexamethasone insert in the upper or lower punctum.
Time Frame: Day 0
Population: Attempts at Upper and Lower insertion
Measure: Count of Participants; unit: Participants
Arm/Group | Lower Punctum Insertion (Group 1) | Upper Punctum Insertion (Group 2)
Number analyzed (Participants) | 39 | 40
Participants
  One Attempt | 38 | 35
  Two Attempts | 1 | 5

ADVERSE EVENTS:
Time Frame: 30 days
Description: An AE is any untoward or unfavorable medical occurrence in a participant, including any abnormal sign, symptom or disease, temporally associated with the participants' participation in the research, whether or not considered related to the participant's participation on the research.
Arm/Group | Lower Punctum Insertion (Group 1) | Upper Punctum Insertion (Group 2)
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/40
Other Adverse Events (participants affected / at risk) | 4/39 | 4/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lower Punctum Insertion (Group 1) (N=39) | Upper Punctum Insertion (Group 2) (N=40)
Increased IOP (Eye disorders) | 0 (0) | 1 (1) — An AE is any untoward or unfavorable medical occurrence in a participant, including any abnormal sign, symptom or disease, temporarily associated with the participants' participation in the research.
CME (Eye disorders) | 1 (1) | 1 (1) — An AE is any untoward or unfavorable medical occurrence in a participant, including any abnormal sign, symptom or disease, temporarily associated with the participants' participation in the research.
Blurred Vision (Eye disorders) | 0 (0) | 1 (1) — An AE is any untoward or unfavorable medical occurrence in a participant, including any abnormal sign, symptom or disease, temporarily associated with the participants' participation in the research.
Anterior Chamber Inflammation (Eye disorders) | 1 (1) | 1 (1) — An AE is any untoward or unfavorable medical occurrence in a participant, including any abnormal sign, symptom or disease, temporarily associated with the participants' participation in the research.
Corneal Edema (Eye disorders) | 1 (1) | 0 (0) — An AE is any untoward or unfavorable medical occurrence in a participant, including any abnormal sign, symptom or disease, temporarily associated with the participants' participation in the research.
Insert Fell Out (Eye disorders) | 1 (1) | 0 (0) — An AE is any untoward or unfavorable medical occurrence in a participant, including any abnormal sign, symptom or disease, temporarily associated with the participants' participation in the research.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-26): https://cdn.clinicaltrials.gov/large-docs/15/NCT05372315/Prot_SAP_000.pdf